CLINICAL TRIAL: NCT05726474
Title: Comparison of the Effect of Two Types of Physical Exercise on the Improvement of Exercise Capacity, Diastolic Function, Endothelial Function, and Arterial Stiffness in Patients With Heart Failure With Preserved Ejection Fraction (ExIC-FEp Study)
Brief Title: Comparison of the Effect of Two Types of Physical Exercises in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: ExIC-FEp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBPLY/21/180501/000112
Record Dates: First submitted 2022-10-20; First posted 2023-02-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Physical Exercise; Exercise Capacity; Diastolic Function; Endothelial Function; Arterial Stiffness
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combined exercise (Experimental)
  Interventions: Behavioral: Combined exercise
- High interval training (Experimental)
  Interventions: Behavioral: High interval training
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Combined exercise — Patients will exercise for 40 minutes three times a week on an ergometric bicycle at 50-60% of VO2max, 60-70% of HRmax, 11-13 on the Borg scale, without ergometer at 50-60% of VO2max, 60-70% of HRmax, 11-13 on the Borg scale, without shortness of breathing difficulty. In addition, strength training will be performed (bench press, leg press, leg curl, leg machine, bench press, leg press, leg curl, leg curl, leg machine). leg curls, leg curls, rowing machine, triceps dips, pectoral pull-ups) twice a week. week. Strength training will be performed with 15 repetitions per exercise and per session, with a corresponding workload of 15 repetitions. session, with a workload corresponding to 60% to 65% of the 1-repetition maximum (1RM) measured at (1RM) measured at the beginning and at the end of the intervention.
  Arms: Combined exercise
Behavioral: High interval training — Patients will perform three training sessions per week. Each training session begins with a 10-minute warm-up at moderate intensity (corresponding to 50-60% of VO2max, 60-70% of HRmax, 11-13 on the Borg scale, no shortness of breath) before cycling, four 4-minute intervals at high intensity (corresponding to 85-90% of VO2max, 90-95% of HRmax, 15-17 on the Borg scale, shortness of breath). Each interval will be separated by 3 minutes of active pauses, with a HRmax of 50-70%. The training session will end with 3 minutes of cool down at moderate intensity (corresponding to 50-60%). moderate intensity (corresponding to 50-60% of VO2max, 60-70% of HRmax, 11-13 on the Borg scale, without difficulty). Borg scale, no shortness of breath). The total exercise time will be 40 minutes for the HIIT group.
  Arms: High interval training

SUMMARY:
Background: Heart failure (HF) is a chronic disease with a very important and increasingly severe social and health impact with a prevalence of 6.8% in Spain. HF with preserved ejection fraction (HFpEF) represents approximately 50% of all patients with HF. In the absence of pharmacological treatments that have succeeded in reducing mortality or morbidity in this pathology, it is recommended that interventions be directed at prevention, symptomatic treatment of HF and treatment of comorbidities to avoid exacerbations, thus physical exercise is recognized as an important adjunct in the treatment of HF and is recommended by the guidelines of the American College of Cardiology (ACC)/American Heart Association (AHA) and the European Society of Cardiology (ESC). Currently, aerobic exercise is the most studied physical exercise in this population, but in recent years high-intensity interval training (HIIT) and the combination of aerobic exercise with strength training (combined exercise) have emerged.

Objectives: The overall objective of this study is to compare the effectiveness of combined training and HIIT on exercise capacity, diastolic function, endothelial function, and arterial stiffness in patients with HFpEF. The specific objectives of this study are: a) to compare the effectiveness of combined training and HIIT on quality of life in patients with HFpEF and b) to analyze the cost-effectiveness of combined training and HIIT versus conventional treatment in patients with HFpEF.

Methodology: The ExIC-FEp study will be a single-blind randomized clinical trial with 3 arms (combined exercise, HIIT and a control group), conducted at the Health and Social Research Center of the University of Castilla-La Mancha, to analyze two types of supervised physical exercise in patients with HFpEF for 6 months. Patients with HFpEF will be randomly assigned (1:1:1) to the combined exercise, HIIT or control group. All participants will be examined, at baseline (prior to randomization), at three months (mid-intervention) and at six months (at the end of the intervention). Participants will undergo physical examination, echocardiography, maximal cardiopulmonary stress test, and measurement of endothelial function and arterial stiffness. In addition, sociodemographic variables, quality of life, physical activity, adherence to the Mediterranean diet, strength, spirometry and blood sampling will be measured.

Expected scientific contributions: this randomized clinical trial will represent a a significant advance in the scientific evidence available on the efficacy of physical exercise in the treatment of HFpEF, through: (a) transfer of the results to physicians, nurses and patients; (b) dissemination of results through scientific articles, doctoral theses and participation in congresses; (c) press releases and press conferences with the aim of disseminating the research results to the population; (d) dissemination through social networks to improve the social impact; and (e) design and content development of a web page.

ELIGIBILITY:
Inclusion Criteria:

1. Heart Failure with preserved ejection fraction picture (diagnosis according to ESC 2021 criteria)

   1. Signs and symptoms of Heart Failure
   2. A left ventricular ejection fraction of ≥50%.
   3. Objective evidence of cardiac structural and/or functional abnormalities consistent with the presence of left ventricular diastolic dysfunction/elevated left ventricular filling pressures, including elevated natriuretic peptides.
2. Sedentary men and women (structured exercise <2 x 30 min/week).
3. Age ≥40 years
4. Written informed consent
5. Clinically stable for 6 weeks
6. Optimal medical treatment for ≥6 weeks

Exclusion Criteria:

1. Non-cardiac causes of heart failure symptoms:

   * Significant valvular or coronary artery disease - Uncontrolled hypertension or arrhythmias.
   * Primary cardiomyopathies
2. Significant pulmonary disease (FEV1<50% predicted, GOLD III-IV)
3. Inability to exercise or conditions that may interfere with exercise intervention.
4. Myocardial infarction in the last 3 months
5. Signs of ischaemia during maximal cardiopulmonary exercise test.
6. Comorbidity that may influence one-year prognosis 7. Participation in another clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Change from Baseline exercise capacity at 3 months
  Maximal cardiopulmonary stress test with Ergoline600 ergometer bicycle.
E velocity | Change from Baseline E velocity at 3 months
  E velocity in m/s
Endothelial function | Change from Baseline endothelial function at 3 months
  Carotid intima-media thickness: by ultrasound with the Sonosite SII device.
Arterial stiffness | Change from Baseline arterial stiffness at 3 months
  Pulse wave velocity and augmentation index
A velocity | Change from Baseline A velocity at 3 months
  A velocity in m/s
E/A ratio | Change from Baseline E/A ratio at 3 months
  E/A ratio
e' velocity | Change from Baseline e' velocity in m/s at 3 months
  e' velocity in m/s
E/e' ratio | Change from Baseline E/e' ratio at 3 months
  E/e' ratio
ejection fraction | Change from Baseline ejection fraction at 3 months
  percentage of ejection fraction
left ventricular volume index | Change from Baseline left ventricular volume index at 3 months
  left ventricular volume index
end-diastolic volume | Change from Baseline end-diastolic volume at 3 months
  end-diastolic volume
left ventricular mass | Change from Baseline left ventricular mass at 3 months
  left ventricular mass
left atrial diameter | Change from Baseline left atrial diameter at 3 months
  left atrial diameter
isovolume relaxation time | Change from Baseline isovolume relaxation time at 3 months
  isovolume relaxation time in seg
deceleration time | Change from Baseline deceleration time at 3 months
  deceleration time in m/s
left atrial volume index | Change from Baseline left atrial volume index at 3 months
  left atrial volume index

SECONDARY OUTCOMES:
Sociodemographic variables | Baseline
  Age, sex and socioeconomic level
Patient's medical history | Baseline
  Comorbidities and medication
Weight | Change from Baseline weight at 3 months
  Weight in kilogram
Muscular strength | Change from Baseline Muscular strength at 3 months
  Handgrip force to be determined with TKK 5401 Grip-D dynamometer.
Spirometry | Change from Baseline spirometry at 3 months
  Forced vital capacity (FVC), forced expiratory volume in the first second (FEV1) and FEV1/FVC ratio.
Glucose | Change from Baseline Glucose at 3 months
  Glucose
Physical activity | Change from Baseline phisical activity at 3 months
  Accelerometry. Time of physical activity
HQoL | Change from Baseline HQoL at 3 months
  Validated 12-item health questionnaire (SF-12). From 0 to 12 (higher values better HQoL)
Adherence to the Mediterranean diet | Change from Baseline Adherence to the Mediterranean diet at 3 months
  Validated 14-item questionnaire on adherence to the Mediterranean diet (MEDAS-14). From 0 to 14 (higher values better Adherence)
height | Change from Baseline height at 3 months
  height in centimeters
BMI | Change from Baseline BMI at 3 months
  BMI in kg/m2
waist circumference | Change from Baseline waist circumference at 3 months
  waist circumference in cm
body fat | Change from Baseline body fat at 3 months
  percentage of body fat
blood pressure | Change from Baseline blood pressure at 3 months
  systolic and diastolic blood pressure in mmHg
total cholesterol | Change from Baseline total cholesterol at 6 months
  total cholesterol
triglycerides | Change from Baseline triglycerides at 6 months
  triglycerides
HDL-cholesterol | Change from Baseline HDL-cholesterol at 6 months
  HDL-cholesterol
LDL-cholesterol | Change from Baseline LDL-cholesterol at 6 months
  LDL-cholesterol
apolipoproteins A1 and B | Change from Baseline apolipoproteins A1 and B at 6 months
  apolipoproteins A1 and B
insulin | Change from Baseline insulin at 6 months
  insulin
ultra-sensitive C-reactive protein | Change from Baseline ultra-sensitive C-reactive protein at 6 months
  ultra-sensitive C-reactive protein
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | Change from Baseline N-terminal pro-B-type natriuretic peptide (NT-proBNP) at 6 months
  N-terminal pro-B-type natriuretic peptide (NT-proBNP)
HbA1c | Change from Baseline HbA1c at 6 months
  HbA1c

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Castulla-La Mancha, Cuenca, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cavero-Redondo I, Saz-Lara A, Bizzozero-Peroni B, Nunez-Martinez L, Diaz-Goni V, Calero-Paniagua I, Matinez-Garcia I, Pascual-Morena C. Accuracy of the 6-Minute Walk Test for Assessing Functional Capacity in Patients With Heart Failure With Preserved Ejection Fraction and Other Chronic Cardiac Pathologies: Results of the ExIC-FEp Trial and a Meta-Analysis. Sports Med Open. 2024 Jun 18;10(1):74. doi: 10.1186/s40798-024-00740-6. PMID 38886304